CLINICAL TRIAL: NCT04300127
Title: Pioglitazone for the Treatment of Idiopathic Gastroparesis (PIOGAS Study)
Brief Title: Pioglitazone for Idiopathic Gastroparesis
Acronym: PIOGAS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00184232
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pioglitazone (Experimental): Candidates who after the screening period are eligible to receive Pioglitazone
  Interventions: Drug: Pioglitazone 30 mg

INTERVENTIONS:
Drug: Pioglitazone 30 mg — Patients will received 30 mg of Pioglitazone once a day for 8 weeks

SUMMARY:
The principal objective of this pilot study will be to evaluate whether 8 weeks of treatment of pioglitazone will improve symptoms as measured by the Gastrointestinal Symptom Index (GCSI) in patients with Idiopathic Gastroparesis.

DETAILED DESCRIPTION:
Objective • The principal objective of this pilot study will be to evaluate whether 8 weeks of treatment of pioglitazone will improve symptoms as measured by the Gastrointestinal Symptom Index Daily Diary (GCSI-DD) in patients with Idiopathic Gastroparesis

Secondary objectives of this study include:

* To determine the effects of pioglitazone on other symptoms associated with gastroparesis using the Patient Assessment of Upper Gastrointestinal Symptom Severity Index (PAGI-SYM) and the Gastrointestinal Symptom Rating Scale (GSRS),
* To determine the effects of pioglitazone on gastric emptying as measured by the 13C- Spirulina breath test,
* To determine the effects of pioglitazone on satiety as measured by a liquid caloric test
* To determine the effects of pioglitazone on depression and anxiety using the Beck Depression Inventory and State-Trait Anxiety Scores,
* To determine the effects of pioglitazone on Quality of Life using the PAGI-QoL and Short Form (SF)-36 questionnaire,
* To determine the effects of pioglitazone on markers of inflammation (CRP and ESR) and serum cytokine levels
* To determine the nature and incidence of adverse effects from a 12-week course of pioglitazone.

Treatment group

• Pioglitazone (30 mg po qd)

Population • Age 18 years or older at registration with nausea, vomiting, and other symptoms suggestive of patients with chronic nausea and vomiting of presumed gastric origin, with symptomatic gastroparesis.

Study duration

* Up to 4 weeks of screening prior to pioglitazone treatment
* 8 weeks of treatment starting at initial dose of pioglitazone
* 4 weeks of washout period
* Length of recruitment: 16 months

Sample size justification

* Total of 23 patients
* Primary comparison: Baseline PAGI-SYM score versus 4, 8, and 12 weeks.

Number of clinical centers

• Johns Hopkins Bayview Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at registration
* Diagnosis of gastroparesis as documented by gastric emptying scintigraphy (4-hour emptying after a low-fat meal with any combination of 2 and 4 hour retention of >60% and 10% respectively)
* Ongoing symptoms referable to gastroparesis (i.e. Nausea and vomiting, bloating, and abdominal pain)
* Exclusion of other causes of symptoms such as mechanical gastrointestinal obstruction, uncontrolled esophagitis, peptic ulcer disease, etc. By standard radiographic or endoscopic tests
* Females will be required to use adequate contraceptive methods during study participation as determined by the Principal Investigator and the study team members

Exclusion Criteria:

* Another active disorder, which could explain symptoms in the opinion of the investigator
* Age < than 18 years
* Pregnancy or nursing
* Previous surgery of the upper gastrointestinal tract, including vagotomy
* Another active disorder, which could explain symptoms in the opinion of the investigator
* Use of narcotics more than 3 days per week
* Significant hepatic injury as defined by significant alanine aminotransferase (ALT) and aspartate aminotransferase (AST) elevations of greater than 2 x upper limit of normal (ULN) or a Child-Pugh score of 10 or greater
* Serious systemic disease, such as recent myocardial infarction/unstable angina, decompensated congestive heart failure, severe pulmonary disease with dyspnea at rest, or altered mental status from any cause
* Diabetes as defined by HbA1c >6.5 and/or fasting blood sugar of >125 mg/DL
* Contraindications to pioglitazone such as hypersensitivity or allergy
* Concurrent use of: estradiol, ethynyl estradiol, mestranol, pazopanib, warfarin, digoxin, atorvastatin, ranitidine, gemfibrozil, fexofenadine, midazolam
* Any other condition, which in the opinion of the investigator would impede compliance or hinder the completion of the study
* History of bladder cancer or family history of bladder cancer
* Failure to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Treisman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone Group: Candidates who are deemed eligible after the screening period will receive Pioglitazone 30 mg once daily for 8 weeks.
Period: Baseline
Arm/Group | Pioglitazone Group
Started | 14
Completed | 14
Not Completed | 0
Period: First Intervention - 4 Weeks Treatment
Arm/Group | Pioglitazone Group
Started | 14
Completed | 12
Not Completed | 2
Period: Second Intervention - 4 Weeks Treatment
Arm/Group | Pioglitazone Group
Started | 12
Completed | 12
Not Completed | 0
Period: Third Intervention - 4 Weeks of Wash Out
Arm/Group | Pioglitazone Group
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pioglitazone
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.31 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Severity of Gastrointestinal Symptoms as Assessed by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index
Description: The effect of Pioglitazone on nausea, early satiety, postprandial fullness, and upper abdominal pain as per changes in patient scoring in The American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index (GCSI) which has been designed to assess symptoms associated with gastroparesis. Symptoms are rated as none (0), mild (1), moderate (2), severe (3), very severe (4) scale of the worst severity of the symptom over the last 24 hours. Values reported represent the mean participant scale choice.
Time Frame: Baseline, later monthly up to 3 months.
Population: Participants who started time point are reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pioglitazone Group
Number analyzed (Participants) | 14
score on a scale
  Baseline | 2.9 (0.9)
  1st month of treatment | 2.3 (1.1)
  2nd month of treatment: number analyzed (Participants) | 12
  2nd month of treatment | 2.2 (1.1)
  3rd month / washout: number analyzed (Participants) | 12
  3rd month / washout | 2.6 (0.8)

2. Secondary Outcome: Patient Assessment of Upper Gastrointestinal Symptom Severity Index (PAGI-SYM)
Description: The Patient Assessment of Gastrointestinal Symptoms (PAGI-SYM) questionnaire is a patient-reported tool designed to evaluate the severity of upper gastrointestinal symptoms across multiple domains, including nausea/vomiting, postprandial fullness/early satiety, bloating, upper abdominal pain, and heartburn/regurgitation. Each symptom is rated on a 0 to 5 Likert scale, where 0 indicates no symptoms and 5 represents very severe symptoms, with higher scores reflecting worse symptom severity. The total PAGI-SYM score is typically calculated as the average of individual domain scores, resulting in a possible score range of 0 to 5. The mean participant scale choice is reported.
Time Frame: Baseline and later monthly up to 3 months
Population: Participants who started time point are reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pioglitazone
Number analyzed (Participants) | 14
score on a scale
  Baseline | 2.6 (0.9)
  1st month of treatment | 1.9 (0.9)
  2nd month of treatment: number analyzed (Participants) | 12
  2nd month of treatment | 1.9 (0.9)
  3rd month / washout: number analyzed (Participants) | 12
  3rd month / washout | 2.3 (0.8)

3. Secondary Outcome: Functional Status as Assessed by the SF-36v2 Health Survey
Description: The effect of Pioglitazone on quality of life assessed by the SF-36v2 Health Survey. The SF-36v2 is a 36-item, self-report measure designed to assess quality of life in patients. This measure also provides two summary scores (physical and mental health) and eight scale scores. The eight sections are: vitality, physical functioning, bodily pain and general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability, i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Baseline, later monthly up to 3 months
Population: Participants who started time point are reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pioglitazone
Number analyzed (Participants) | 14
score on a scale
  Physical Functioning - Baseline | 54.3 (17.6)
  Physical Functioning - 1st month | 64.6 (20.0)
  Physical Functioning - 2nd month: number analyzed (Participants) | 12
  Physical Functioning - 2nd month | 67.1 (24.1)
  Physical Functioning - Washout: number analyzed (Participants) | 12
  Physical Functioning - Washout | 64.6 (22.1)
  Role limitations due to physical activity - Baseline | 40.2 (18.6)
  Role limitations due to physical activity - 1st month | 51.3 (23.2)
  Role limitations due to physical activity - 2nd month: number analyzed (Participants) | 12
  Role limitations due to physical activity - 2nd month | 60.4 (27.2)
  Role limitations due to physical activity - 3rd month / Washout: number analyzed (Participants) | 12
  Role limitations due to physical activity - 3rd month / Washout | 47.2 (30.9)
  Role limitations due to emotional problems - Baseline | 65.5 (29.9)
  Role limitations due to emotional problems - 1st month | 68.5 (30.3)
  Role limitations due to emotional problems - 2nd month: number analyzed (Participants) | 12
  Role limitations due to emotional problems - 2nd month | 77.8 (25.5)
  Role limitations due to emotional problems - 3rd month / Washout: number analyzed (Participants) | 12
  Role limitations due to emotional problems - 3rd month / Washout | 68.9 (30.9)
  Pain - Baseline | 62.9 (19.3)
  Pain - 1st month | 45.2 (23.7)
  Pain - 2nd month: number analyzed (Participants) | 12
  Pain - 2nd month | 41.7 (21.3)
  Pain - 3rd month/Washout: number analyzed (Participants) | 12
  Pain - 3rd month/Washout | 48.5 (23.9)
  Emotional well being - Baseline | 46 (8.1)
  Emotional well being - 1st month | 45.7 (20.4)
  Emotional well being - 2nd month: number analyzed (Participants) | 12
  Emotional well being - 2nd month | 48.7 (9.8)
  Emotional well being - 3rd month / Washout: number analyzed (Participants) | 12
  Emotional well being - 3rd month / Washout | 46.9 (11)
  Energy / fatigue - Baseline | 35.7 (7.3)
  Energy / fatigue - 1st month | 33.6 (17.4)
  Energy / fatigue - 2nd month: number analyzed (Participants) | 12
  Energy / fatigue - 2nd month | 35.4 (9.2)
  Energy / fatigue - 3rd month / Washout: number analyzed (Participants) | 12
  Energy / fatigue - 3rd month / Washout | 35.5 (7.6)
  Social functioning - Baseline | 51.8 (6.7)
  Social functioning - 1st month | 48.2 (6.7)
  Social functioning - 2nd month: number analyzed (Participants) | 12
  Social functioning - 2nd month | 52.1 (8.9)
  Social functioning - 3rd month / Washout: number analyzed (Participants) | 12
  Social functioning - 3rd month / Washout | 50 (5.6)
  General health - Baseline | 63.6 (9.1)
  General health - 1st month | 55.7 (20.7)
  General health - 2nd month: number analyzed (Participants) | 12
  General health - 2nd month | 60.8 (10.6)
  General health - 3rd month / Washout: number analyzed (Participants) | 12
  General health - 3rd month / Washout | 63.2 (7.2)

4. Secondary Outcome: C- Reactive Protein Level in Blood
Description: The effect of Pioglitazone on Inflammatory markers as per changes in the values of C reactive protein (CRP) in blood. Normal CRP levels are below 3.0 mg/L.
Time Frame: Baseline and 2 months after treatment initiation.
Population: Participants who started time point are reported
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pioglitazone
Number analyzed (Participants) | 14
mg/L
  Baseline CRP | 2.5 (3.9)
  8 weeks CRP: number analyzed (Participants) | 12
  8 weeks CRP | 5.1 (12.1)

5. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: The effect of Pioglitazone on Inflammatory markers as per changes Erythrocyte Sedimentation Rate (ESR) in blood. Results are reported as the millimeters of clear fluid (plasma) that are present at the top portion of the tube after one hour. The normal range is 0 to 22 mm/hr for men and 0 to 29 mm/hr for women. Values above these ranges are considered worse.
Time Frame: Baseline and 2 months after treatment initiation
Population: Participants who started time point are reported
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Pioglitazone
Number analyzed (Participants) | 14
mm/h
  Baseline ESR | 14.5 (20.3)
  2 Months ESR: number analyzed (Participants) | 12
  2 Months ESR | 14.8 (13.1)

6. Secondary Outcome: Mood as Assessed by the Beck Depression Inventory
Description: The effect of Pioglitazone on mood as per changes in the score of Beck Depression Inventory (BDI-II). The BDI-II is a commonly used, reliable 21-item self-report measure designed to assess for depression. Individuals are asked to respond to each question based on a two-week time period. The BDI-II is widely used as an indicator of the severity of depression, but not as a diagnostic tool. BDI-II items are rated on a 4-point scale ranging from 0 to 3 based on the severity of each item. The maximum total score range is 0-63. Higher total scores indicate more severe depressive symptoms.
Time Frame: Baseline, later monthly up to 3 months
Population: Participants who started time point are reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pioglitazone
Number analyzed (Participants) | 14
score on a scale
  Baseline BDI-II | 17.9 (11.8)
  4 Weeks BDI-II | 8.6 (8.2)
  8 Weeks BDI-II: number analyzed (Participants) | 12
  8 Weeks BDI-II | 8.8 (7.4)
  Washout BDI-II: number analyzed (Participants) | 12
  Washout BDI-II | 12.6 (9.4)

7. Secondary Outcome: Mood as Assessed by the State-Trait Anxiety Inventory
Description: The effect of Pioglitazone on mood as per changes in the score of the State-Trait Anxiety Inventory (STAI). The STAI is a 40-item self-report measure designed to assess anxiety. This measure provides two subscale scores (State and Trait). STAI is one of the first tests to assess both state and trait anxiety separately. Each type of anxiety has its own scale of 20 different questions that are scored. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Time Frame: Baseline, later monthly up to 3 months
Population: Participants who started time point are reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pioglitazone
Number analyzed (Participants) | 14
score on a scale
  State Anxiety - Baseline | 44.1 (12.8)
  State Anxiety - 1st month | 35.8 (13.9)
  State Anxiety - 2nd month: number analyzed (Participants) | 12
  State Anxiety - 2nd month | 38.7 (15)
  State Anxiety - 3rd month / Washout: number analyzed (Participants) | 12
  State Anxiety - 3rd month / Washout | 36.8 (18.2)
  Trait Anxiety - Baseline | 43.3 (14.2)
  Trait Anxiety - 1st month | 33.9 (15.6)
  Trait Anxiety - 2nd month: number analyzed (Participants) | 12
  Trait Anxiety - 2nd month | 38.4 (11.2)
  Trait Anxiety - 3rd month / Washout: number analyzed (Participants) | 12
  Trait Anxiety - 3rd month / Washout | 39.7 (13)

ADVERSE EVENTS:
Time Frame: Up to 3.5 months
Arm/Group | Pioglitazone
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=14)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Leucopenia (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Headaches (Nervous system disorders) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1)
Vomit (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT04300127/Prot_SAP_000.pdf